CLINICAL TRIAL: NCT06904378
Title: Phase I/II Clinical Trial of Ontegimod and Gemcitabine/Nab-paclitaxel as Second Line Therapy for Metastatic Pancreatic Ductal Adenocarcinoma: Reprogramming Tumor-associated Myeloid Cells
Brief Title: Ontegimod and Gemcitabine/Nab-paclitaxel as Second Line Therapy for Metastatic Pancreatic Ductal Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 25-x095; P50CA272213 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic cancer CD11b; Gemcitabine
MeSH Terms: interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Sequential for Phase I portion of trial and parallel for Phase II portion of trial. Participants will be randomized 6:1 to the experimental arm (Ontegimod/gemcitabine/nab-paclitaxel) vs the control arm (gemcitabine/nab-paclitaxel alone) in the Phase II portion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I Dose de-escalation (starting dose): Ontegimod + Gemcitabine + Nab-paclitaxel (Experimental): Ontegimod is an oral medication taken twice daily on Days 1-21 of each 28-day cycle. The starting dose is 800 mg. Gemcitabine and nab-paclitaxel will be given as per standard of care (intravenous on Days 1, 8, and 15 of each 28-day cycle).
  Interventions: Drug: Ontegimod; Drug: Gemcitabine; Drug: Nab paclitaxel
- Phase 2 Experimental Arm: Ontegimod + Gemcitabine + Nab-paclitaxel (Experimental): Ontegimod is an oral medication taken twice daily on Days 1-21 of each 28-day cycle. The dose will determined during the Phase I portion of the trial. Gemcitabine and nab-paclitaxel will be given as per standard of care (intravenous on Days 1, 8, and 15 of each 28-day cycle).
  Interventions: Drug: Ontegimod; Drug: Gemcitabine; Drug: Nab paclitaxel
- Phase 2 Control Arm: Gemcitabine + Nab-paclitaxel (Active Comparator): Gemcitabine and nab-paclitaxel will be given as per standard of care (intravenous on Days 1, 8, and 15 of each 28-day cycle).
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Ontegimod — Per assigned dose level.
  Arms: Phase 2 Experimental Arm: Ontegimod + Gemcitabine + Nab-paclitaxel; Phase I Dose de-escalation (starting dose): Ontegimod + Gemcitabine + Nab-paclitaxel
Drug: Gemcitabine — The dose of gemcitabine is 1000 mg/m^2.
  Other Names: Gemzar
Drug: Nab paclitaxel — The dose of nab-paclitaxel is 125 mg/m^2.
  Other Names: Abraxane

SUMMARY:
The investigators hypothesize that CD11b agonism reprograms the tumor microenvironment (TME) to overcome resistance to checkpoint immunotherapy in pancreatic ductal adenocarcinoma (PDAC). Therefore, the investigators propose an open label phase I/II clinical trial of Ontegimod with gemcitabine and nab-paclitaxel in unresectable pancreatic ductal adenocarcinoma prior to future studies incorporating anti-PD1 checkpoint immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas.
* Measurable or evaluable disease per RECIST 1.1.
* Lesions amenable to research biopsy, if biopsy is deemed safe and low risk.
* Previously treated with first-line systemic therapy for unresectable/advanced or metastatic PDAC and experienced progression or became intolerant to the therapy and is in need of another line of systemic therapy in the opinion of the investigator.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN, unless there are liver metastases in which case AST and ALT ≤ 5.0 x IULN
  * Creatinine ≤ 1.5 x IULN or Creatinine clearance > 50 mL/min by Cockcroft-Gault
* The effects of Ontegimod on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 120 days after last dose of Ontegimod or 180 days after last dose of nab-paclitaxel/gemcitabine. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Received more than one line of treatment or received gemcitabine or nab-paclitaxel in the metastatic setting. Prior therapy in the adjuvant or neoadjuvant therapy will count as a line of treatment if progression occurred less than 6 months after the last dose of systemic therapy. The following exception applies:

  * If treated in the adjuvant or neoadjuvant setting with systemic therapy and progression occurred greater than 6 months after last dose, the adjuvant or neoadjuvant systemic therapy may have included gemcitabine or nab-paclitaxel. If progression occurred within 6 months of the last dose of systemic therapy in the adjuvant or neoadjuvant setting, then that therapy must not have included gemcitabine or nab-paclitaxel.
* Current use or anticipated need for alternative, holistic, naturopathic, or botanical formulations used for the purpose of cancer treatment.
* Major surgery (defined as surgery that requires general anesthesia) within 28 days of anticipated start date of Ontegimod.
* Chemotherapy, small molecular directed therapy, and/or radiation therapy within 14 days of anticipated start date of Ontegimod.
* History of other malignancy with the exception of 1) malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease and 2) known indolent malignancies that do not require treatment and will likely not alter the course of treatment of metastatic PDAC.
* History of allogeneic organ or stem cell transplant.
* Currently receiving any other investigational agents.
* Patients with known, untreated brain metastases. Patients with treated brain metastases are allowed if post-treatment brain-imaging after CNS-directed therapy shows no evidence of progression.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to Ontegimod, gemcitabine, nab-paclitaxel, or other agents used in the study.
* Average QTc (Bazett) >470 msec on screening EKG.
* Gastrointestinal condition which could prevent absorption of Ontegimod, or inability to digest Ontegimod.
* Clinically significant peripheral neuropathy grade 2 or worse.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test within 7 days of C1D1.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussing with the Principal Investigator.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of C1D1 except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted. Inhaled intranasal, intra-articular, and topical steroid uses are permitted.
* Patients with known Gilbert's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) (Phase I only) | After completion of cycle 1 (each cycle is 28 day) for all Phase I participants (estimated to be 12 months)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. In the absence of excess toxicity, the maximum tolerated dose will become the recommended phase 2 dose (RP2D).
Number of participants with dose-limiting toxicities (DLTs) (Phase I only) | After completion of cycle 1 (each cycle is 28 day)
  DLTs are defined in the protocol.
Progression-free rate at 6 months (RP2D participants in Phase I and Phase II participants only) | At 6 months from start of treatment

SECONDARY OUTCOMES:
Frequency of adverse events (RP2D participants in Phase I and Phase II participants in experimental arm only) | From start of treatment through 30 days after last dose of treatment (estimated to be 7 months)
  - The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Objective response rate (ORR) (RP2D participants in Phase I and Phase II participants in experimental arm only) | Through completion of treatment (estimated to be 6 months)
  * ORR is defined as the proportion of patients with disease control (Complete response + Partial response).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) (RP2D participants in Phase I and Phase II participants in experimental arm only) | Through completion of follow-up (estimated to be 18 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall survival (OS) (RP2D participants in Phase I and Phase II participants in experimental arm only) | Through completion of follow-up (estimated to be 18 months)
  OS is defined as the duration of time from start of treatment to time of death from any cause. The alive patients are censored at last follow-up date.
Disease control rate (DCR) (RP2D participants in Phase I and Phase II participants in experimental arm only) | Through completion of follow-up (estimated to be 18 months)
  * DCR is defined as the proportion of patients with disease control (Complete response + Partial response + Stable Disease) per RECIST 1.1.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Grierson, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu